CLINICAL TRIAL: NCT06253988
Title: Evaluating the Effect of a Mixture of Lactobacillus Brevis and Lactobacillus Plantarum on the Management of Periodontitis Stage III Grade C Molar-incisor Pattern in Egyptian Patients ( Randomize Control Trial)
Brief Title: Effect of Probiotics on Periodontitis Stage III Grade C Molar-incisor Pattern
Acronym: RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Shaymaa Hussein Rafat Kotb, Assistant lecturere of oral medicine ,periodontology departement at sphinx university, Sphinx university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AUAREC202300010-2
Record Dates: First submitted 2024-01-09; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis; Agg. actinomycetemcomitans; JP2 genotype; PCR; local delivery drug; probiotics
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: Sixty-five patients having periodontitis stage III grade C molar-incisor pattern. Screening for A. actinomycetemcomians (A.a) and the JP2 genotype was done using conventional polymerase chain reaction (PCR). Patients positive for (A. a) were randomly divided into two groups. Group I: received conventional periodontal treatment combined with topically applied probiotic, while Group II: received conventional periodontal treatment only. Both groups were evaluated microbiologically and clinically.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group probiotic (Active Comparator): received conventional periodontal treatment combined with topically applied probiotic
  Interventions: Drug: Probiotic Formula
- Group placebo (Placebo Comparator): received conventional periodontal treatment only.
  Interventions: Drug: placebo formula

INTERVENTIONS:
Drug: Probiotic Formula — intra-pocket formula (local delivery drug)
  Other Names: A mixture of Lactobacillus brevis and Lactobacillus plantarum
  Arms: Group probiotic
Drug: placebo formula — intra-pocket formula (local delivery drug)
  Other Names: placebo
  Arms: Group placebo

SUMMARY:
the research highlight the effectiveness of probiotics as adjuncts to SRP in the treatment of periodontitis stage III grade C molar-incisor pattern

DETAILED DESCRIPTION:
Background data : Periodontitis is a common disease that represents a public health problem. Aggregatibacter actinomycetemcomitans (A. a ) especially the JP2 genotype plays a major role in the pathogenesis of periodontitis. The aim of this study is to evaluate the effect of topically applied probiotics on the management of periodontitis stage III grade C molar-incisor pattern.

Methods: Sixty-five patients having periodontitis stage III grade C molar-incisor pattern. Screening for A. actinomycetemcomians (A.a) and the JP2 genotype was done using conventional polymerase chain reaction (PCR). Patients positive for (A. a) were randomly divided into two groups. Group I: received conventional periodontal treatment combined with topically applied probiotic, while Group II: received conventional periodontal treatment only. Both groups were evaluated microbiologically and clinically. Quantitative assessment of A. a levels was done by real time PCR (qPCR) at baseline as well as one week, 4 weeks, and 12 weeks after treatment. Clinical parameters were assessed before treatment as well as 3,6 and 9 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients have periodontitis stage III grade C molar-incisor pattern .

Exclusion Criteria:

* Pregnant or nursing women,
* smokers,
* patients received periodontal therapy,
* systemic antimicrobials or anti-inflammatory drugs in the last six
* patients with unacceptable oral hygiene

Ages: 10 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
quantitative assessment of A. actinomycetemcomians levels by picogram | at baseline (before treatment) used by conventional PCR
  Microbiological evaluation by picogram
Assessment of clinical periodontal parameter : Probing pocket Depth (PPD) by mm | at base line , 1 , 3 , 6 months
  Clinical evaluation mm
Assessment of clinical periodontal parameter : Clinical Attachment Level (CAL) by mm | at base line , 1 , 3 , 6 months
  Clinical evaluation by "mm"

SECONDARY OUTCOMES:
quantitative assessment of A. actinomycetemcomians levels by picogram | baseline ,1 ,3 and 6 months
  microbiological by picogram

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim H Ibrahim, Ass.prof., Principal Investigator — Al-Azhar University; Mohamed A EL-Mokhtar, Prof, Study Director — Assiut University; Mohamed F Edrees, prof., Principal Investigator — Al-Azhar University; Heba A Hammad, Ass.prof, Study Director — Assiut University
Locations (1):
- Alazhar university ,faculty of Dental Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Effect of probiotics on periodontitis stage III grade C molar-incisor pattern
Supporting Information: SAP
Time Frame: 1 month
Access Criteria: DOI: 10.21203/rs.3.rs-3837892/v1
URL: https://doi.org/10.21203/rs.3.rs-3837892/v1

REFERENCES:
- See also: Orchid — https://orcid.org/my-orcid?orcid=0000-0002-8404-438X
- See also: National library of Medicine — https://www.ncbi.nlm.nih.gov/myncbi/collections/mybibliography/
- See also: web of science — http://www.webofscience.com/wos/author/record/ABE-1539-2022